CLINICAL TRIAL: NCT04231227
Title: Validity and Reliability of the Turkish Version of Test of Arm Selective Control and the Relationship Between Upper Limb Selective Motor Control and Motor Functions in Children With Cerebral Palsy
Brief Title: The Validity and Reliability of the Turkish Version of TASC and the Relationship Between SMC and Motor Functions
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Seyma Kilcioglu, M.Sc. Student, Gazi University
Other Study IDs: Upper Limb SMC in CP
Record Dates: First submitted 2020-01-10; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy, Spastic; Cerebral Palsy; Cerebral Palsy Spastic Diplegia; Cerebral Palsy Quadriplegic; Cerebral Palsy, Monoplegic
Keywords: cerebral palsy; selective motor control; upper limb; upper limb functions; gross motor functions
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Selective motor control (SMC) impairment in children with cerebral palsy (CP) includes movement patterns dominated by flexor or extensor synergy affecting functional movements. The research was designed to investigate the validity and the reliability of the Turkish version of the Test of Arm Selective Control (TASC) (which is improved to evaluate SMC in children with spastic CP) and in order to provide more understanding of the relationship between SMC and upper extremity and gross motor functions. The study included 21 hemiplegic, 11 diplegic and 4 quadriplegic children with CP whose ages are 4 to 18 years and Gross Motor Function Classification System (GMFCS) level changes from 1 to 4, and their parents. In order to evaluate the gross motor function of children, GMFCS and the ability to hold objects with their hands in daily activities were evaluated with Manual Ability Classification System (MACS). ABILHAND-Kids scale was applied to evaluate upper extremity performance. TASC scale was used to evaluate the upper extremity SMC of children.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of spastic CP
* being able to understand the commands required for the test,
* being between the ages of 3-18,
* being GMFCS level I to IV.

Exclusion Criteria: • Having undergone orthopedic surgery or Botulinum Toxin A (BTX-A) within the last 6 months

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children in Special Education Centers
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Test of Arm Selective Control | from July to September 2018
  an upper limb selective motor control evaluation tool.
Abilhand- Kids Questionnaire | from July to September 2018
  to assess a child's unimanual and bimanual upper limb activities
Manual Ability Classification System | from July to September 2018
  to assess manual abilities of children
Gross Motor Function Classification System | from July to September 2018
  To assess gross motor functions of children

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)